CLINICAL TRIAL: NCT00669630
Title: The GoodNEWS (Genes, Nutrition, Exercise, Wellness, and Spiritual Growth) Trial
Brief Title: The GoodNEWS Lifestyle Enhancement Program
Acronym: GoodNEWS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01HL087768 (NIH); R01HL087768-01 (NIH)
Record Dates: First submitted 2008-04-28; First posted 2008-04-30 (Estimated); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Cardiovascular Disease; Hypertension; Diabetes; Obesity
Keywords: Community-based Participatory Research (CBPR); Vulnerable population; High-risk population; African-Americans; Health Disparities; Clinical Trial
MeSH Terms: conditions — Cardiovascular Diseases; Hypertension; Diabetes Mellitus; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Lay Health Promoter (LHP) with maintenance — Lay Health Promoters (LHPs) and their congregations will join an existing social and organizational support network, comprised of LHPs and congregations who are part of an active community health improvement collaborative.
  Other Names: Faith-Based Intervention; Faith-Based Program

SUMMARY:
This study will train Lay Health Promoters (LHPs) from African-American churches to administer healthy living lessons and activities to their congregations in order to improve overall health and address cardiovascular disease. The primary hypothesis is that LHP training combined with a well supported maintenance strategy will be more effective than LHP training alone in reducing risk factors for cardiovascular disease.

DETAILED DESCRIPTION:
The GoodNEWS Trial is an 18-month effectiveness trial with an 18-month extended maintenance study, among 20 African-American and low-income congregations participating in the GoodNEWS faith-based lay health promotion program. After training, congregations will be randomized to either GoodNEWS with a health maintenance intervention (GoodNEWS-I) or GoodNEWS program alone (GoodNEWS-PA). The maintenance intervention combines elements of the medical care model and features of community-based support. Primary data collection will occur at baseline, 18, and 36 months with the two primary outcomes being levels of physical activity as measured by 7- Day Physical Activity Recall (PAR) and dietary change as measured by the Diet History Questionnaire (DHQ). The primary hypothesis is that the maintenance group will significantly increase physical activity and healthy eating behavior compared to the program only group. We also hypothesize that lipoprotein and glucose levels, and blood pressure will be significantly improved over baseline in the GoodNEWS-I group and that these changes will be significantly greater than in the GoodNEWS-PA group. At the end of the trial, both groups will continue in an 18-month extended maintenance study.

ELIGIBILITY:
Inclusion Criteria:

* Member of selected church congregations in the predominantly African-American geographical area of Dallas, Texas, known as South Dallas or the Southern Sector.
* Between the ages of 18 -70 years

Exclusion Criteria:

* Anyone under the age of 18
* Anyone who is not an active member of one of the participating churches

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 392 (Actual)
Dates: Start 2008-09 (Actual); Primary Completion 2011-09 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Diet History Questionnaire; 7 - Day Physical Activity Recall | Baseline, 18 months, and 36 months

SECONDARY OUTCOMES:
Blood pressure; Total cholesterol, HDL, LDL, Triglycerides; Glucose level; Hemoglobin A1C (Diabetics only) | Baseline, 18-months, and 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Mark J. DeHaven, Ph.D., Principal Investigator — UT Southwestern Medical Center at Dallas
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

REFERENCES:
- [Derived] Carson JA, Michalsky L, Latson B, Banks K, Tong L, Gimpel N, Lee JJ, Dehaven MJ. The cardiovascular health of urban African Americans: diet-related results from the Genes, Nutrition, Exercise, Wellness, and Spiritual Growth (GoodNEWS) trial. J Acad Nutr Diet. 2012 Nov;112(11):1852-8. doi: 10.1016/j.jand.2012.06.357. Epub 2012 Sep 18. PMID 22995059